CLINICAL TRIAL: NCT04046419
Title: Turkish Validity and Reliability of "Health Care Providers and Impairment Relationship Scale (HC-PAIRS)"
Brief Title: In Turkish Version "Health Care Providers and Impairment Relationship Scale (HC-PAIRS)"
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Saracoglu, PhD, Pt., Kutahya Health Sciences University
Other Study IDs: KutahyaMSUt
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2021-03

CONDITIONS: Chronic Low-back Pain; Health Personnel Attitude
Keywords: validity, reliability, Turkish version, HC-PAIRS

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Turkish validity and reliability — 1. Explanation of the Turkish version of the scale.
  2. Translating the Turkish version of the scale into English to ensure consistency with the original scale.
  3. First application of scales to participants.
  4. Second application of the scales to the participants.
  5. Statistical analysis and scaling

SUMMARY:
The aim of this study was to determine the Turkish validity and reliability of ''Health Care Providers and Impairment Relationship Scale HC (HC-PAIRS)'' developed by Dr Rainville.

DETAILED DESCRIPTION:
Low back pain is one of the reasons for applying to health institutions. Low back pain, which seriously affects patients' lives and leads to major financial losses, causes serious deficiencies in both developing and developed countries. Health professionals' perception of pain, factors associated with pain and fear avoidance attitudes of patients affect the success of treatment. The aim of this study is to determine the Turkish version, validity and reliability of ''Health Care Providers and Impairment Relationship Scale (HC-PAIRS)''. 165 physiotherapist working with chronic low back pain were included in the study. In order to determine the reliability of the scale, the intraclass correlation coefficient (ICC) will be used to determine the level of the relationship between the results of the first and second measurements. Cronbach's alpha coefficient will be used for homogeneity of the questions in the scale. For concurrent validity, correlation coefficient will be used to determine the agreement between the previously validated scales and the Turkish version of HC PAIRS.

ELIGIBILITY:
Inclusion Criteria:

* Graduate with a bachelor's degree in physiotherapy and rehabilitation
* To have worked in patients with chronic low back pain

Exclusion Criteria:

* Not having experience in the clinic about low back pain

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out by physiotherapists working in the KSBU Evliya Celebi Hospital or accessible via internet.
Sampling Method: Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
The Health Care Providers' Pain and Impairment Relationship Scale | 10 minute
  The Health Care Providers' Pain and Impairment Relationship Scale (HC-PAIRS) is a questionnaire for assessing the attitudes and beliefs of health care providers about functional expectations for CLBP patients.17 It consists of 15 statements rated on a 6-point Likert scale ranging from "totally disagree" to "totally agree."
Turkish version of Tampa Scale for Kinesiophobia | 10 minute
  TSK was used for the assessment of kinesiophobia. The items are rated on a 4-point Likert-type scale (1=definitely disagree, 4=completely agree) and the total score is between 17 and 68 points. Higher total score indicates higher level of kinesiophobia.

SECONDARY OUTCOMES:
Pain Attitudes and Beliefs Scale for Physiotherapists (PABS-PT) | 10 minute.
  This tool was developed to distinguish between biomedical and biopsychosocial orientations toward the treatment of low back pain in physiotherapists. The scale uses a 6-point Likert-type scale (1=definitely disagree, 6=definitely agree). Treatment orientation is measured on the biomedical (factor 1) and biopsychosocial (factor 2) subscales. Subscale scores are calculated by simply adding the scores corresponding to the selected response for each item. The subscale with the highest score indicates the respondent's dominant treatment orientation

CONTACTS AND LOCATIONS:
Overall Officials: Cihan C AKSOY, PhD, Study Director — Kutahya Health Science University; İsmail SARACOGLU, PhD, Principal Investigator — Kutahya Health Science University; Lütfiye AKKURT, MSc, Principal Investigator — Kutahya Health Science University
Locations (1):
- Kutahya Health Science University, Kütahya, Turkey (Türkiye)